CLINICAL TRIAL: NCT00658931
Title: Cymbalta for Depression as a Complication of Bereavement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jefferson Clinic, P.C. (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: John L. Shuster, Jr., MD, Jefferson Clinic, PC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIJ-US-X047
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Depression; Bereavement
Keywords: Depression; Bereavement; Pilot Projects; Antidepressant Drugs
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Drug treatment with Cymbalta

INTERVENTIONS:
Drug: Drug treatment with Cymbalta — Drug treatment with Cymbalta
  Other Names: Duloxetine Hydrochloride

SUMMARY:
The primary objective of this pilot project is to evaluate the efficacy of Cymbalta for bereavement-associated depression. Participating patients will be treated with Cymbalta in doses up to 60mg daily for eight (8) weeks. The primary outcome measure for this study will be the 17-item Hamilton Rating Scale for Depression (HRSD-17). In pursuit of this objective, we will test the following hypothesis: After eight weeks of open-label treatment with Cymbalta for bereavement-associated depression, at least half of the participants will achieve remission, as measured by a score of 7 or less on the HRSD-17.

Secondary objectives of this project are:

* To determine the tolerability of Cymbalta treatment among patients with bereavement-associated depression (as measured by adverse events and the proportion of participants who discontinue Cymbalta before completing eight weeks of study treatment);
* To determine the effect of Cymbalta treatment on grief in patients with bereavement-associated depression (as measured by the Texas Revised Inventory of Grief and the Inventory of Complicated Grief after eight weeks of treatment compared to baseline); and
* To determine the effect of Cymbalta treatment on health status, pain, and other co-morbid symptoms in patients with bereavement-associated depression (as measured by the Edmonton Symptom Assessment System and the Medical Outcomes Study 12-item Short Form Health Survey administered at Weeks 2, 4, and 8 and compared to baseline).

DETAILED DESCRIPTION:
The primary objective of this pilot project is to evaluate the efficacy of Cymbalta for bereavement-associated depression. Participating patients will be treated with Cymbalta in doses up to 60mg daily for eight (8) weeks. The primary outcome measure for this study will be the 17-item Hamilton Rating Scale for Depression (HRSD-17). In pursuit of this objective, we will test the following hypothesis: After eight weeks of open-label treatment with Cymbalta for bereavement-associated depression, at least half of the participants will achieve remission, as measured by a score of 7 or less on the HRSD-17.

Secondary objectives of this project are:

* To determine the tolerability of Cymbalta treatment among patients with bereavement-associated depression (as measured by adverse events and the proportion of participants who discontinue Cymbalta before completing eight weeks of study treatment);
* To determine the effect of Cymbalta treatment on grief in patients with bereavement-associated depression (as measured by the Texas Revised Inventory of Grief and the Inventory of Complicated Grief after eight weeks of treatment compared to baseline); and
* To determine the effect of Cymbalta treatment on health status, pain, and other co-morbid symptoms in patients with bereavement-associated depression (as measured by the Edmonton Symptom Assessment System and the Medical Outcomes Study 12-item Short Form Health Survey administered at Weeks 2, 4, and 8 and compared to baseline).

This pilot study is an eight-week, open-label clinical antidepressant treatment trial using Cymbalta (duloxetine hydrochloride) in doses between 20mg and 60mg daily for patients with co-morbid depression and bereavement. Twenty (20) patients who have sustained the loss of a first-degree relative (spouse, child, parent, or sibling) within the past two years AND meet criteria for a major depressive episode at the time of screening will be recruited for participation in this study. Patients who tolerate and respond to Cymbalta treatment will be offered maintenance therapy with Cymbalta for up to one year at the effective dose. We expect that Cymbalta treatment will be associated with substantial remission and response rates, as measured by HRSD-17 scores. Similarly, we expect substantial mean reductions in measures of grief and bereavement, with improvements in measures of pain, symptom burden, and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Must have sustained the loss of a first-degree relative (spouse, partner, child, parent, sibling, or person otherwise described by the patient as a first-degree relative) within the past two years and one of the two following features must also be present:

  1. at least two months must have passed since the death prior to enrollment in the study, OR
  2. there must be evidence of marked functional impairment (as defined in the DSM-IV description of Bereavement, v62.82);
* Must meet criteria for a major depressive episode as defined in DSM-IV;
* Onset of this depressive episode must have occurred after the death of the first-degree relative (if the relative's death was unexpected) OR no more then three months prior to the death of the relative (if the relative's death was expected);
* HRSD-17 score of >17 at baseline assessment;
* Must be in stable medical health;
* Must be able to communicate in English; AND
* Must be willing and able to travel to the Cooper Green Mercy Hospital or the Jefferson Clinic, PC for evaluations according to the study protocol.

Exclusion Criteria:

* History of Dysthymic Disorder or a depressive episode preceding the death of the first-degree relative by more than three months;
* History or symptoms of mania or psychosis (e.g., bipolar disorders, schizophrenia and other psychotic disorders);
* Evidence of current alcohol or other substance abuse or dependence;
* Evidence of clinically significant dementia or cognitive impairment (from history or a score on the screening Mini Mental State Exam of 23 or less);
* Concomitant use of other antidepressants (patients can be enrolled after taper and clearance of other antidepressant medications);
* Concomitant use of medications known to have potential for clinically significant interaction with Cymbalta (patients can be enrolled after taper and clearance of other medications, if other medications can be safely discontinued).
* Suicidal thoughts with intent or plan, or other situations where the patient is judged to be a high risk of suicide;
* Known hypersensitivity to Cymbalta or any of its inactive ingredients;
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization or potential need to use an MAOI during the study or within 5 days of discontinuation of study drug; OR
* Any of the following medical conditions present:

  1. Hepatic impairment or insufficiency,
  2. Hyponatremia,
  3. Narrow-angle glaucoma,
  4. History of seizures,
  5. Unstable hypertension, OR
  6. Pregnancy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
17-item Hamilton Rating Scale for Depression (HRSD-17) | Eight weeks

SECONDARY OUTCOMES:
Texas Revised Inventory of Grief (TRIG) | Eight weeks
Prolonged Grief Disorder (PG-13) Measure | Eight weeks
Clinical Global Impressions - Severity of Illness (CGI-S) | Eight weeks
Clinical Global Impressions - Improvement (CGI-I) | Eight weeks
Mini-Mental State Examination (MMSE) | Eight weeks
Edmonton Symptom Assessment System (ESAS) | Eight weeks
Medical Outcomes Study 12-item Short Form Health Survey (SF-12v2): | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: John L Shuster, MD, Principal Investigator — Jefferson Clinic, PC
Locations (1):
- Jefferson Clinic, PC, Birmingham, Alabama, United States